CLINICAL TRIAL: NCT03883152
Title: Yeur-Hur Lai, PhD, RN, School of Nursing, College of Medicine, National Taiwan University
Brief Title: Eating Difficulties in HNC Patients - Influencing Factors and Short and Long Term Impacts on PF and Depression
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201703066RIND
Record Dates: First submitted 2018-12-03; First posted 2019-03-20 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2019-12

CONDITIONS: Head and Neck Cancer
Keywords: Eating Difficulties; Chewing; Swallowing; Head and neck cancer; Depression; Physical function; Nutrition
MeSH Terms: conditions — Head and Neck Neoplasms; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Head and neck cancer: Eating difficulty is one of the most common problems for head and neck cancer (HNC), in particular, who are in advanced disease stage and receive surgery, radiation (RT) or concurrent radio-chemotherapy (CCRT) (Vissink, Burlage, Spijkervet, Jansma, & Coppes, 2003; Lazarus et al., 2014). The consequences of multi-treatment bring structural and functional changes in oral, pharynx, or larynx and influence the normal eating process (Logemann et al., 2006; Lazarus et al., 2013; Patterson, McColl, Wilson, Carding, Rapley, 2015; McLaughlin, 2014).

SUMMARY:
Background: Eating difficulty is one of the most common problems faced by head and neck cancer (HNC) patients and it might influence patients' general function and psychological function. Unfortunately, the eating difficulties in HNC patients are not fully understood due to limited research presented.

Purposes: The study is a 2-year longitudinal following up research. The purpose of the study aim to (1) examine the characteristics and severity of eating difficulty, (2) identify factors related to the eating difficulty, and (3) short and long-term impact and correlation of eating difficulty on HNC patients' general physical condition and depression.

Method: Eligible patient will be HNC patients receiving surgery and CCRT. Patients will be recruited and assessed in 6 time points: before first CCRT (T1) and 4weeks, 8 week, 12 week , 6 month, and 12 month from CCRT (T2~T6). Patients will be assessed nutrition status, body weight, fatigue severity, and grip power of the dominant hand, and depression. IRB and patient consents will be obtained before data collection. The descriptive and correlational analyses will be applied to analyze the data. The investigators plan to recruit 125 subjects. The longitudinal data will be analyzed by GEE to examine the changes of main variables and predictors of eating difficulty.

Expected Outcome: The results of this study will provide evidence about HNC patients' eating difficulty. It will increase health care professionals' understanding about HNC patients' problems in eating difficulties, related factors and their relationship with general function. The investigators hope to further develop an intervention based on the results to enhance HNC patients' eating function.

DETAILED DESCRIPTION:
This is a longitudinal study which aims to examine the short- and long-term eating difficulties, its related factors and its impacts. The participants will be recruited in the outpatient department of Ear, Nose, and Throat (ENT) in NTUH. The inclusion criteria are (a) diagnosed as head and neck cancer; (b) will be received cancer treatments including surgery and CCRT; (c) age is 20 or older. The exclusion criteria are (a) the patient is inserted a plastic tube, e.g. nasogastric tube (NG) or percutaneous endoscopic gastrostomy tube (PEG), for feeding; (b) patients could not understand the content of questionnaires. The investigators will recruit 100 subjects with complete 12-month data. Concerning 25% patients loss rate, the investigators will recruit 125 subjects at the beginning of the first year.

Patients will be assessed by Chewing Swallowing Inventory (CSI), Mini Nutritional Assessment (MNA), Depression subscale of Hospital Anxiety and Depression Scale (HADS), Symptom Severity Scale (SSS), 0-10 general Fatigue severity numerical scale, and disease and treatment background Information Form (BIF). Grip power of dominant hand will be assessed by hand dynamometer.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with head and neck cancer
* patients with concurrent chemo-radiotherapy (CCRT)

Exclusion Criteria:

* primary unknown
* conscious unclear
* recurrence or with bone meta

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eating difficulty is one of the most common problems for head and neck cancer (HNC), in particular, who are in advanced disease stage and receive surgery, radiation (RT) or concurrent radio-chemotherapy (CCRT) (Kendall, 2008; Vissink, Burlage, Spijkervet, Jansma, & Coppes, 2003; Lazarus, Husaini, Hu,…et al., 2014). The consequences of multi-treatment bring structural and functional changes in oral, pharynx, or larynx and influence the normal eating process (Logemann et al., 2006; Lazarus CL, Husaini H, Anand,…et al., 2013; Patterson, McColl, Wilson, Carding, Rapley, 2015; McLaughlin, 2014).
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
Change in the Chewing Swallowing Inventory (CSI) | Patients will be recruited and assessed in 6 time points: before first CCRT (T1) and 4weeks, 8 week, 12 week , 6 month, and 12 month from CCRT (T2~T6).
  This questionnaire is used to assess HNC patients' eating difficulties. CSI is a 21-item 5-point Likert's scale. The items represent the alteration of oral mucus, intake condition (abilities to chew, opening mouth, smelling, tasting, and tongue movement, and time spending for intake), and assistance for maintaining patients' independence. The score range of CSI is from 0 to 84. The higher score indicates the more severe difficulty of swallowing and intake. After revised the CSI content regarding the responses from 30 head-and-neck cancer patients, twenty-one items in the CSI were selected if the Index of Content Validity (CVI) were 0.86 or higher, and Cronbach's alpha was 0.91.
Change in The Mini Nutritional Assessment (MNA) | Patients will be recruited and assessed in 6 time points: before first CCRT (T1) and 4weeks, 8 week, 12 week , 6 month, and 12 month from CCRT (T2~T6).
  MNA is a validated tool consisted of nutrition screening and general assessment to early detect the malnourished geriatric patients who are age at 65 and older (Guigoz, Vellas, & Garry, 1996). The total score of the MNA is 30. The cut-off point to distinguish the elder's nutrition was in three types: a) MNA ≥ 24 indicating an adequate nutritional status, b) MNA between 17 and 23.5 indicating a risk of malnutrition, and c) MNA < 17 indicating protein-calorie malnutrition. With these cut points, sensitivity was found to be 96%, specificity 98%, and predictive value 97% (Vella, Guigoz, & Garry, et al, 1999). Satisfactory reliability and validity of the MNA-Chinese version has been validated to assess nutrition for the elder in Taiwan (Tsai, Ho, & Chang, 2008; Tsai, Change, Wang, & Liao, 2010), and to assess nutrition of patients with liver cancer (Hsu, Tsai, Chan, Wang, & Chung, 2012; Tsai, Hsu, Chan, & Chang, 2011).
Change in the Depression Subscale of Hospital Anxiety and Depression Scale (HADS-D) | Patients will be recruited and assessed in 6 time points: before first CCRT (T1) and 4weeks, 8 week, 12 week , 6 month, and 12 month from CCRT (T2~T6).
  We will use 14-item HADS to assess patients' anxiety and depression (Zigmond & Snaith, 1983). The HADS has 7 items that measure anxiety and 7 that measure depression. The total score of each subscale is ranged from 0 to 21 with a higher score indicating a higher level of anxiety and depression. The Taiwanese version of HADS has been developed and validated showed promising psychometrics (Chen et al., 2010; Cheng, Hao, Lin, & Yeh, 2000).
Change in the Symptom Severity Scale (SSS) | Patients will be recruited and assessed in 6 time points: before first CCRT (T1) and 4weeks, 8 week, 12 week , 6 month, and 12 month from CCRT (T2~T6).
  Patients' symptom severity was measured by the Symptom Severity Scale, and that was developed and modified to determine treatment-related symptoms in head and neck cancer patients (Chen et al., 2010). The 20-item SSS contains items related to swallowing difficulty, eating difficulty, oral mucositis, speech difficulty, fatigue, poor appetite, pain, cough, apnea, constipation, diarrhea, nausea, and vomiting. Each item is rated on an 11-point scale of 0 to 10, with 0 indicating "no such symptom at all" and 10 indicating "extreme severity of the symptom." The SSS has been demonstrated to be a reliable scale in oral cancer-related studies in Taiwan, with Cronbach's alpha coefficients ranging from 0.82 to 0.91 (Chen et al., 2010; Chen et al., 2013).
Change in the Background Information Form | Patients will be recruited and assessed in 6 time points: before first CCRT (T1) and 4weeks, 8 week, 12 week , 6 month, and 12 month from CCRT (T2~T6).
  Background Information Form displays participants' characteristics. Patients' demographics describe age, sex, and marital status. Patients' clinical characteristics, which are categorical variables, show cancer diagnoses, stages, recurrence, categories and time of treatments for HNC cancer, and reconstruction within surgery.
Change in the Hand Dynamometer Evaluation | Patients will be recruited and assessed in 6 time points: before first CCRT (T1) and 4weeks, 8 week, 12 week , 6 month, and 12 month from CCRT (T2~T6).
  We will use the hand dynamometer to assess HNC patients' hands' grip power. It will represent the general energy level of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Yeur-Hur Lai, Professor, Study Chair — School of Nursing, College of Medicine, National Taiwan University
Locations (1):
- Yeur-Hur Lai, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guigoz Y, Vellas B, Garry PJ. Assessing the nutritional status of the elderly: The Mini Nutritional Assessment as part of the geriatric evaluation. Nutr Rev. 1996 Jan;54(1 Pt 2):S59-65. doi: 10.1111/j.1753-4887.1996.tb03793.x. No abstract available. PMID 8919685
- [Background] Vellas B, Guigoz Y, Garry PJ, Nourhashemi F, Bennahum D, Lauque S, Albarede JL. The Mini Nutritional Assessment (MNA) and its use in grading the nutritional state of elderly patients. Nutrition. 1999 Feb;15(2):116-22. doi: 10.1016/s0899-9007(98)00171-3. PMID 9990575
- [Background] Tsai AC, Ho CS, Chang MC. Assessing the prevalence of malnutrition with the Mini Nutritional Assessment (MNA) in a nationally representative sample of elderly Taiwanese. J Nutr Health Aging. 2008 Apr;12(4):239-43. doi: 10.1007/BF02982628. PMID 18373032
- [Background] Tsai AC, Chang TL, Wang YC, Liao CY. Population-specific short-form mini nutritional assessment with body mass index or calf circumference can predict risk of malnutrition in community-living or institutionalized elderly people in taiwan. J Am Diet Assoc. 2010 Sep;110(9):1328-34. doi: 10.1016/j.jada.2010.06.003. PMID 20800124
- [Background] Tsai AC, Hsu WC, Chan SC, Chang TL. Usefulness of the mini nutritional assessment in predicting the nutritional status of patients with liver cancer in Taiwan. Nutr Cancer. 2011;63(3):334-41. doi: 10.1080/01635581.2011.535966. PMID 21462083
- [Background] Hsu WC, Tsai AC, Chan SC, Wang PM, Chung NN. Mini-nutritional assessment predicts functional status and quality of life of patients with hepatocellular carcinoma in Taiwan. Nutr Cancer. 2012;64(4):543-9. doi: 10.1080/01635581.2012.675620. Epub 2012 Apr 20. PMID 22519878
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Herrmann C. International experiences with the Hospital Anxiety and Depression Scale--a review of validation data and clinical results. J Psychosom Res. 1997 Jan;42(1):17-41. doi: 10.1016/s0022-3999(96)00216-4. PMID 9055211
- [Background] Lloyd-Williams M, Friedman T, Rudd N. An analysis of the validity of the Hospital Anxiety and Depression scale as a screening tool in patients with advanced metastatic cancer. J Pain Symptom Manage. 2001 Dec;22(6):990-6. doi: 10.1016/s0885-3924(01)00358-x. PMID 11738161
- [Background] Chen ML, Chang HK, Yeh CH. Anxiety and depression in Taiwanese cancer patients with and without pain. J Adv Nurs. 2000 Oct;32(4):944-51. PMID 11095234
- [Background] Chen SC, Lai YH, Liao CT, Lin CC. Psychometric testing of the Impact of Event Scale-Chinese Version (IES-C) in oral cancer patients in Taiwan. Support Care Cancer. 2005 Jul;13(7):485-92. doi: 10.1007/s00520-005-0775-x. Epub 2005 Feb 17. PMID 15717159
- [Background] Chen SC, Lai YH, Liao CT, Lin CC, Chang JT. Changes of symptoms and depression in oral cavity cancer patients receiving radiation therapy. Oral Oncol. 2010 Jul;46(7):509-13. doi: 10.1016/j.oraloncology.2010.02.024. Epub 2010 Mar 21. PMID 20308004
- [Background] Chen SC, Lai YH, Liao CT, Chang JT, Lin CY, Fan KH, Huang BS. Supportive care needs in newly diagnosed oral cavity cancer patients receiving radiation therapy. Psychooncology. 2013 Jun;22(6):1220-8. doi: 10.1002/pon.3126. Epub 2012 Jun 25. PMID 22730021
- [Background] Vissink A, Burlage FR, Spijkervet FK, Jansma J, Coppes RP. Prevention and treatment of the consequences of head and neck radiotherapy. Crit Rev Oral Biol Med. 2003;14(3):213-25. doi: 10.1177/154411130301400306. PMID 12799324
- [Background] Lazarus CL, Husaini H, Hu K, Culliney B, Li Z, Urken M, Jacobson A, Persky M, Tran T, Concert C, Palacios D, Metcalfe-Klaw R, Kumar M, Bennett B, Harrison L. Functional outcomes and quality of life after chemoradiotherapy: baseline and 3 and 6 months post-treatment. Dysphagia. 2014 Jun;29(3):365-75. doi: 10.1007/s00455-014-9519-8. Epub 2014 Mar 8. PMID 24609609
- [Background] Lazarus CL, Husaini H, Anand SM, Jacobson AS, Mojica JK, Buchbinder D, Urken ML. Tongue strength as a predictor of functional outcomes and quality of life after tongue cancer surgery. Ann Otol Rhinol Laryngol. 2013 Jun;122(6):386-97. doi: 10.1177/000348941312200608. PMID 23837392
- [Background] Logemann JA, Rademaker AW, Pauloski BR, Lazarus CL, Mittal BB, Brockstein B, MacCracken E, Haraf DJ, Vokes EE, Newman LA, Liu D. Site of disease and treatment protocol as correlates of swallowing function in patients with head and neck cancer treated with chemoradiation. Head Neck. 2006 Jan;28(1):64-73. doi: 10.1002/hed.20299. PMID 16302193
- [Background] Patterson JM, McColl E, Wilson J, Carding P, Rapley T. Head and neck cancer patients' perceptions of swallowing following chemoradiotherapy. Support Care Cancer. 2015 Dec;23(12):3531-8. doi: 10.1007/s00520-015-2715-8. Epub 2015 Apr 8. PMID 25851803
- [Background] McLaughlin L. Taste dysfunction and eating behaviors in survivors of head and neck cancer treatment. Medsurg Nurs. 2014 May-Jun;23(3):165-70, 184. PMID 25137792